CLINICAL TRIAL: NCT04910841
Title: Feasibility of Using the "CGM GUARDIAN 2" Interstitial Fluid Glucose Measurement System in Intensive Care Medicine
Acronym: GALI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-AOI-10
Record Dates: First submitted 2021-05-27; First posted 2021-06-02 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-08

CONDITIONS: Hyperglycemia; Hypotension; Shock, Septic
MeSH Terms: conditions — Hyperglycemia; Hypotension; Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Connect (Experimental)
  Interventions: Device: CGM GUARDIAN 2

INTERVENTIONS:
Device: CGM GUARDIAN 2 — continuous blood glucose monitoring system

SUMMARY:
Glycemic imbalances are very common in shock patients admitted to intensive care units. A blood glucose control every 2 hours is routinely performed in patients requiring insulin therapy. In practice, we use a protocol and management software called "CPG" (Personalized Control of Blood Glucose). This involves taking capillary samples from the fingertips. In addition to the pain generated, local haematomas and sensitivity disorders have been described. Night-time sampling also leads to repeated awakenings. The "CGM GUARDIAN 2" system has been validated for the measurement of glucose in interstitial fluid in insulin-dependent diabetic patients. An electrode is placed on the patient's abdomen or arm for up to 6 days. This electrode consists of a needle that is inserted subcutaneously only during the placement. The sugar level is read using a sensor placed on the electrode and an insulin pump (which will not deliver therapy (for our study) and which will be used only as an information reader to know the glucose level and trends). Interstitial fluid is automatically drawn from the electrode every minute and averaged every 5 minutes.

This device has not yet been validated in resuscitation patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient in septic shock
* Arterial hypotension requiring noradrenaline
* Hyperglycaemia requiring insulin therapy

Exclusion Criteria:

* Patients under guardianship, curatorship or deprived of liberty
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Glucose level | Day 6

CONTACTS AND LOCATIONS:
Overall Officials: Florent BILGER, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No